CLINICAL TRIAL: NCT07059195
Title: Non-Invasive Techniques to Maintain Neck Flexion and Reduce Anastomotic Tension After Tracheal Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Talal Mahomud, Assisstent lecturer at cardiothorathic department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-6--2MD
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Maintain Neck Flexion and Reduce Anastomotic Tension After Tracheal Resection
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group A (Non-invasive group) (Active Comparator): Patients in this group will have postoperative cervical spine flexion maintained using non-invasive techniques, such as a cervical collar or cervical-thoracic orthosis.
  Interventions: Procedure: cervical collar or cervical-thoracic orthosis.
- • Group B (Conventional group) (Active Comparator): Patients in this group will have cervical spine flexion maintained using traditional chin-to-chest (Grillo) suturing
  Interventions: Device: chin-to-chest (Grillo) suturing

INTERVENTIONS:
Procedure: cervical collar or cervical-thoracic orthosis. — postoperative cervical spine flexion maintained using non-invasive techniques, such as a cervical collar or cervical-thoracic orthosis.
  Arms: • Group A (Non-invasive group)
Device: chin-to-chest (Grillo) suturing — cervical spine flexion maintained using traditional chin-to-chest (Grillo) suturing
  Arms: • Group B (Conventional group)

SUMMARY:
Tracheal surgery represents a relatively recent advancement in the field of thoracic surgery. The trachea has unique anatomical and physiological challenges that historically rendered surgical manipulation both risky and limited. Early interventions involving the trachea were primarily restricted to emergency tracheostomy procedures, typically performed as life-saving measures during acute airway obstruction (1). Attempts at tracheal reconstruction were largely unsuccessful due to the absence of suitable anesthesia, inadequate surgical tools, and the prevailing belief that tracheal cartilage lacked sufficient regenerative. As a result, tracheal resection and reconstruction were long considered unfeasible (2).

The modern era of tracheal surgery began to take shape in the mid-20th century. While early attempts at tracheal resection were performed with limited success, it was the pioneering work of Dr. Hermes C. Grillo in the 1960s that truly transformed the field. Through systematic study of tracheal anatomy, vascular supply, and biomechanics, Dr. Grillo developed standardized and safe techniques for segmental tracheal resection followed by primary end-to-end anastomosis. His work demonstrated that segmental resection of the trachea followed by primary end-to-end anastomosis was feasible and safe (3)(4).

ELIGIBILITY:
Inclusion Criteria:

* All pediatric and adult patients undergoing tracheal and cricotracheal resection for benign air way stenosis
* All pediatric and adult patients undergoing tracheal and cricotracheal resection for malignant pathologies

Exclusion Criteria:

* patients with previous cervical spine surgery.
* Congenital or acquired spinal deformities.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
cervical spine flexion | 2 years
  Maintain Neck Flexion and Reduce Anastomotic Tension After Tracheal Resection

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided